CLINICAL TRIAL: NCT03823859
Title: Metabolomics of Thyroid Hormones
Acronym: MATcH
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2018-01961
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Central Hypothyroidism; Hypothyroidism; Hyperthyroidism
Keywords: Hypothyroidism; Metabolomics; Thyroid Hormones; Hyperthyroidism
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism | interventions — Absorptiometry, Photon; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: * Blood sampling (fT3, fT4, TSH, Lipids, Glucose, HbA1c)
  * Indirect calorimetry
  * Dual energy X-ray Absorptiometry (DXA)
  Interventions: Diagnostic Test: Indirect calorimetry; Diagnostic Test: Dual energy X-ray Absorptiometry (DXA); Diagnostic Test: Blood sampling
- Patients with thyroid dysfunction: Patients with Primary hypothyroidism newly diagnosed, Primary hypothyroidism substituted, hyperthyroidism, secondary hypothyroidism
  * Blood sampling (fT3, fT4, TSH, Lipids, Glucose, HbA1c)
  * Indirect calorimetry
  * Dual energy X-ray Absorptiometry (DXA)
  Interventions: Diagnostic Test: Indirect calorimetry; Diagnostic Test: Dual energy X-ray Absorptiometry (DXA); Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Indirect calorimetry — Resting energy expenditure
Diagnostic Test: Dual energy X-ray Absorptiometry (DXA) — Body composition
Diagnostic Test: Blood sampling — fT4, fT3, TSH, HDL, LDL, triglycerides, cholesterol, HbA1c, Glucose Thyroid panel

SUMMARY:
The aim of this study is to develop a metabolome signature of thyroid hormone status. The metabolome signature could be useful in diagnosis and treatment of thyroid dysfunction diseases, especially in cases where TSH cannot be reliably used.

DETAILED DESCRIPTION:
Primary Hypothyroidism is a frequent endocrine disorder, where the thyroid gland does not produce sufficient amounts of thyroid hormones. The substitution therapy is guided by measurement of the pituitary gland hormone thyrotropin (TSH). Patients with central hypothyroidism in whom pituitary insufficiency leads to hypothyroidism, TSH cannot be used to guide therapy. So far there are no reliable methods for therapy control in patients with central hypothyroidism.

The measurement of small endogenous metabolites might give investigators a metabolomics profile. This could help to discriminate between euthyroid, hypothyroid and hyperthyroid state and therefore could be used for diagnosis and therapy control of thyroid dysfunction diseases.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Age 18 to 80 years
* BMI 19 to 35 kg/m2
* Informed consent as documented by signature

A) Patients with primary hyperthyroidism TSH < 0.2 mIU/l and free thyroxine (fT4) > 25 pM or fT3 > 8 pM

B) Patients with primary hypothyroidism, currently not sufficiently substituted TSH > 8 milli-International unit (mIU)/l or fT4 < 10 pM

C) Patients with diagnosis of primary hypothyroidism, sufficiently substituted Documented diagnosis of primary hypothyroidism Substitution with L-Thyroxin TSH in target range between 0.5 and 2.5 mIU/l

D) Patients with secondary hypothyroidism Pituitary disease with documented secondary hypothyroidism

Exclusion Criteria:

* Diabetes mellitus (HbA1c >6.5%)
* Severe concomitant diseases: chronic heart failure, liver cirrhosis, kidney failure, active cancer
* Abuse of alcohol or illicit drugs
* Women who are pregnant or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited by means of advertisements (online or in the newspaper).
  Patients will be recruited from the endocrinology outpatient clinics of the Department of Endocrinology, Diabetes and Metabolism, University Hospital Basel and patients referred from practicing endocrinologists.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Metabolome signature of thyroid Hormone Status (MSTH) | baseline/single visit
  The MSTH will be tested against the current standard of diagnosis which is serum TSH level by multiple linear regression.

SECONDARY OUTCOMES:
Resting energy expenditure (REE) | baseline/single visit
  Comparison of REE of healthy volunteers and Patients with thyroid dysfunction, measured by indirect calorimetry.
Body composition concerning muscle mass | baseline/single visit
  Comparison of muscle mass of healthy volunteers and patients with thyroid dysfunction, measured by DXA
Body composition concerning fat mass | baseline/single visit
  Comparison of fat mass of healthy volunteers and patients with thyroid dysfunction, measured by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Betz, PD Dr. med., Study Director — Klinik Endokrinologie, Diabetes und Metabolismus
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland